CLINICAL TRIAL: NCT02085018
Title: A Randomised, Placebo-controlled Trial of Omeprazole in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Pilot Trial Of Omeprazole in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: PPIPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IAFIPF001; 2013-003301-26 (EudraCT Number); IPFPSG12-7 (Other Grant/Funding Number: British Lung Foundation); 13/YH/0284 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-02-09; First posted 2014-03-12 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: omeprazole, idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Experimental): Omeprazole 20 milligrams twice a day taken for 90 days
  Interventions: Drug: Omeprazole
- Matched placebo (Placebo Comparator): Matched placebo twice a day taken for 90 days
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: Omeprazole — Drug
  Other Names: Losec
  Arms: Omeprazole
Drug: Matched placebo — Matched placebo
  Arms: Matched placebo

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a disease of unknown cause in which areas of normal lung tissue are replaced by scars. As a result it becomes harder for the lungs to extract oxygen from the air. IPF is commonly progressive, and around 50% of patients diagnosed with the disease die after approximately 3 years. The most common, troublesome symptoms of IPF are breathlessness on exertion, and cough. No drug treatments have been unequivocally shown to improve the death rate, or to significantly impact upon symptoms, in IPF.

In recent years it has been recognised that cough can be caused by small amounts of liquid coming up from the stomach and "going down the wrong way" into the lungs, a process commonly known as "reflux". As liquid in the stomach is usually acidic, patients' lungs may repeatedly be exposed to small amounts of acid. Reflux is unusually common in IPF and could potentially contribute to the debilitating cough found with the disease. However there are many potential causes for cough in IPF.

Stomach acid can be efficiently "switched off" by drugs called "proton pump inhibitors", one of which is called omeprazole. If reflux of stomach acid does contribute to cough in IPF, omeprazole might be expected to reduce cough. The purpose of this study is therefore to test whether omeprazole does reduce cough in patients with IPF. Sixty patients with IPF will be randomly allocated to have 3 months of omeprazole or a placebo. Neither the patient nor the doctor will be aware which treatment has been given, ie this is a randomised "double-blind", placebo--controlled trial. Patients' cough frequency will be measured before and after treatment and the change in cough frequency compared in those receiving omeprazole and those receiving placebo. Change in cough frequency is the main thing we aim to compare, but a range of other measurements will be assessed such as the numbers of patients eligible to take part, agreeing to randomisation and providing outcome data, patients' lung function, symptom scores, the amount of reflux, and the amount of inflammation in the lungs.

ELIGIBILITY:
Inclusion Criteria:

* IPF is considered the most likely diagnosis by the Regional Interstitial Lung Disease Multidisciplinary Team meeting (ILD-MDT).
* History of cough, with or without exertional dyspnoea.
* High resolution computed tomography (HRCT) scan features of honeycombing in a predominantly basal subpleural distribution.
* Bibasal crackles on auscultation.
* Features of a restrictive ventilatory defect [vital capacity (VC) <90% predicted and/or diffusion factor for carbon monoxide (Tco) <90% predicted].
* Aged 40-85 years.
* Patients taking short courses (eg. 2 months) of proton pump inhibitors (PPI) will be eligible once the treatment has been discontinued for a minimum of 1 month.

Exclusion Criteria:

* Known allergy to Omeprazole or other proton pump inhibitor.
* Concomitant use of warfarin, diazepam, phenytoin, ketoconazole.
* Concomitant use of a regular PPI, antacid, prokinetic or raft alginate during the trial period.
* History of upper respiratory tract infection, lower respiratory tract infection or exacerbation of IPF in the 4 weeks before starting study drugs.
* Active trial of treatment for IPF 9eg. prednisolone, pirfenidone, N-acetylcysteine) started in the 4 weeks before starting study drugs.
* Documented history of hepatic cirrhosis.
* Pregnancy or lactation.
* ILD-MDT considers the most likely cause of he patient's ILD to be a condition other than IPF (eg. rheumatoid lung, systemic sclerosis ILD, asbestosis, chronic hypersensitivity pneumonitis, sarcoidosis, etc.).
* Concurrent enrolment in a trial of a Clinical Trial of Investigational Medicinal Product (CTIMP) for IPF.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
objectively measured cough frequency | 90 days
  the change in frequency of objectively measured cough from beginning of the study to the end of treatment (within 2 weeks of completion of treatment). This will be compared in the two groups.

SECONDARY OUTCOMES:
symptoms of cough | 90 days
  change in symptoms of cough at the end of treatment as measured by validated cough questionnaire
reflux symptoms | 90 days
  change in symptoms of reflux as measured by validated questionnaires
acid and non-acid reflux | 90 days
  change in acid and non-acid reflux measured by oesophageal physiological study
vital capacity (VC) & transfer factor for carbon monoxide (Tco) | 90 days
  change in VC and Tco as measured by lung function tests
6 minute walk distance | 90 days
  change in 6 minute walk distance from baseline to 90 days
assess amount of inflammation in lung | 90 days
  assess markers of lung inflammation in bronchoalveolar lavage (BAL) fluid (eg. concentration of transforming growth factor beta, interleukin-8 etc.)
lung infection rate | 90 days
  assess bronchoalveolar lavage (BAL) fluid for infections over period from baseline to 90 days, also patient reported infection in adverse event diary
adverse events rate | 90 days
  patient reported adverse events, assess lung infection rate in bronchoalveolar fluids over period from baseline to 90 days

OTHER OUTCOMES:
rate of recruitment | 18 months
  Number of participants eligible and consented for study
rate of study completion | 18 months
  Number of participants completing all study procedures (over 90 days for each participant)

CONTACTS AND LOCATIONS:
Overall Officials: John Simpson, FRCP, Study Director — Newcastle University; Ian Forrest, MRCP, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (1):
- The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne & Wear, United Kingdom